CLINICAL TRIAL: NCT04148950
Title: Effects of Compression Stockings and Kinesio Taping Method on Pain, Edema, Functional Capacity and Quality of Life in Patients With Chronic Venous Disease
Brief Title: Effects of Kinesio Taping Method on Functional Capacity and Quality of Life in Patients With Chronic Venous Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Baha Naci, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E.50.0.05.00/17
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Varicose Veins of Lower Limb; Varicose Veins and Edema of Leg; Chronic Venous Hypertension Peripheral; Spider Veins; Telangiectasia
Keywords: Chronic Venous Disease; Kinesio Taping; Compression Stockings; Pain; Edema; Functional Capacity
MeSH Terms: conditions — Varicose Veins; Telangiectasis; Pain; Edema | interventions — Athletic Tape; Stockings, Compression; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping (Experimental): Kinesio Taping group consisted of 29 patients with CVD. Kinesio Taping was applied once a week for a period of 4 weeks. Closed Fan and Closed Basketweave techniques were applied according to the clinical manifestations, intensity of symptoms, and the needs for the areas to be taped. Basketweave technique was used generally for the thigh, and the areas rich in lymph nodes while closed fan technique was used for cruris, and regions of less severe venous reflux or obstruction. Kinesio Taping was slowly removed by the patient 4 days after the application to prevent any allergic reactions. In addition, patients were given calf muscle pump exercises, flexibility exercises, diaphragmatic breathing exercises, and lower extremity elevation.
  Interventions: Other: Kinesio Tape; Other: Exercise Program
- Compression Stockings (Active Comparator): Compression stockings group consisted of 29 patients with CVD. Patients were recommended medium pressure (23-32 mmHg) compression stockings by the physician. Knee high or thigh high compression stockings were given according to the level of symptoms and signs. In addition, patients were given calf muscle pump exercises, flexibility exercises, diaphragmatic breathing exercises, and lower extremity elevation.
  Interventions: Other: Compression Stockings; Other: Exercise Program

INTERVENTIONS:
Other: Kinesio Tape
  Other Names: Medical Adhesive Tape
  Arms: Kinesio Taping
Other: Compression Stockings
  Other Names: Elastic Compression Stockings
  Arms: Compression Stockings
Other: Exercise Program

SUMMARY:
The purpose of this randomised and controlled study is to investigate the effects of Kinesio Taping method and compression stockings, combined with exercise therapy, on pain, edema, functional capacity and quality of life in patients with chronic venous disease. Therefore, the study compares effectiveness of these two methods for chronic venous disease.

DETAILED DESCRIPTION:
Chronic venous disease (CVD), an important cause of morbidity, is one of the most commonly reported chronic medical conditions. Venous hypertension in the lower limbs caused by venous reflux, venous obstruction or calf muscle pump failure is the main pathophysiological mechanism of CVD. The incidence of varicose veins in population varies with geographic region, age, gender and risk factors. The prevalence of trunk varicose veins has been reported 25.9% in women and 12.9% in men. Symptoms include leg pain, edema, pruritus, discomfort, trophic skin changes, venous ulcerations. Reduced quality of life, and limited activities of daily living have been reported due to the symptoms in patients with CVD.

Compression therapies play a major role in the treatment of CVD. Elastic compression stockings reduces residual volume fraction by promoting calf muscle pump function and reducing venous reflux. Periodic contractions of the gastrocnemius muscle has also beneficial impacts on improving calf muscle pump function and reducing venous stasis.

Kinesio Taping, developed by Dr. Kenzo Kase, is a taping method applied for supporting muscle function, correcting joint misalignment, improving lymph and blood flow, decreasing pain and edema. Kinesio Taping increases cutaneous and subcutaneous area by lifting the skin, thus improves movement and circulation. Mixed Kinesio Taping-compression model has been reported to improve venous symptoms, peripheral venous flow, disease severity and quality of life in patients with mild CVD.

Studies comparing conservative treatment techniques and investigating functional capacity in patients with CVD are very limited despite the high prevalence of disease. Therefore, the investigators planned this study to examine the effects of Kinesio Taping method and compression stockings on pain, edema, functional capacity and quality of lifein patients with CVD.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary chronic venous disease after Doppler Ultrasonographic assessment by the physician
* Presence of clinical symptoms of chronic venous disease
* Patients with C1 (telangiectasias, reticular veins), C2 (varicose veins) or C3 (edema) clinical classes of CEAP (clinical, etiologic, anatomic, pathophysiologic) classification system
* Patients not using medication for the treatment of chronic venous disease
* No prior varicose vein surgery
* Being volunteer for participating in the research
* Signing the written informed consent form prior to participation in the study

Exclusion Criteria:

* Deep Vein Thrombosis
* Thrombophlebitis
* Active or healed venous ulcerations
* Hyperpigmentation
* Bleeding varicose veins
* Open wounds and acute infections
* Acute decompensated heart failure
* Uncontrolled hypertension
* Severe cognitive impairment
* Patients with poor adherence to the treatment program
* Allergic reaction to polyacrylate forms of medical adhesives
* Pregnancy

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Pain at 4 weeks | Baseline and week 4
  Intensity of pain was evaluated using the Visual Analogue Scale (VAS). VAS ranges from 0 mm indicating "no pain" to 100 mm indicating "the worst pain possible".

SECONDARY OUTCOMES:
Change from Baseline Edema at 4 weeks | Baseline and week 4
  Peripheral edema was assesed in both lower limbs by using circumference measurement in four areas, including the ankle joint, the knee joint, the widest region of the calf and the widest region of the thigh.
  A flexible, inelastic, 7 mm-wide tape measure with a sensitivity degree of 0.1 cm was used for the measurements.
Change from Baseline Functional Capacity at 4 weeks | Baseline and week 4
  Exercise capacity was measured with the 6 Minute Walk Test (6MWT) according to the ATS guidelines. The 6 minutes wallking distance (6MWD) was recorded in meters. Higher scores indicate a better outcome.
Change From Baseline Short Form-36 at Week 4 | Baseline and week 4
  Short Form-36 [SF-36] (0-100) was performed to assess generic quality of life (QOL). SF-36 consists of 36 items and 8 subscales. These subscales are physical functioning, role functioning physical, bodily pain, general health perception, vitality, social functioning, role functioning emotional, and mental health. The eight subscales are also summarized into mental component summary and physical component summary scores. Mental component summary contains the subscores of vitality, social functioning, role-emotional, and mental health. Physical component summary contains the subscores of physical functioning, role-physical, bodily pain, and general health. All the scores range from 0 to 100. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Baha Naci, PT, MSc, Principal Investigator — Istanbul University - Cerrahpasa; Semiramis Ozyilmaz, Assoc. Prof., Study Director — Bezmialem Vakif University; Zerrin Yigit, MD, Prof., Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Institute of Cardiology, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Beebe-Dimmer JL, Pfeifer JR, Engle JS, Schottenfeld D. The epidemiology of chronic venous insufficiency and varicose veins. Ann Epidemiol. 2005 Mar;15(3):175-84. doi: 10.1016/j.annepidem.2004.05.015. PMID 15723761
- [Background] Piazza G. Varicose veins. Circulation. 2014 Aug 12;130(7):582-7. doi: 10.1161/CIRCULATIONAHA.113.008331. No abstract available. PMID 25114187
- [Background] Coon WW, Willis PW 3rd, Keller JB. Venous thromboembolism and other venous disease in the Tecumseh community health study. Circulation. 1973 Oct;48(4):839-46. doi: 10.1161/01.cir.48.4.839. No abstract available. PMID 4744789
- [Background] Bartholomew JR, King T, Sahgal A, Vidimos AT. Varicose veins: newer, better treatments available. Cleve Clin J Med. 2005 Apr;72(4):312-4, 319-21, 325-8. doi: 10.3949/ccjm.72.4.312. PMID 15850243
- [Background] Cools AM, Witvrouw EE, Danneels LA, Cambier DC. Does taping influence electromyographic muscle activity in the scapular rotators in healthy shoulders? Man Ther. 2002 Aug;7(3):154-62. doi: 10.1054/math.2002.0464. PMID 12372312
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Result] Ibegbuna V, Delis KT, Nicolaides AN, Aina O. Effect of elastic compression stockings on venous hemodynamics during walking. J Vasc Surg. 2003 Feb;37(2):420-5. doi: 10.1067/mva.2003.104. PMID 12563216
- [Result] Orsted HL, Radke L, Gorst R. The impact of musculoskeletal changes on the dynamics of the calf muscle pump. Ostomy Wound Manage. 2001 Oct;47(10):18-24. PMID 11890075
- [Result] Aguilar-Ferrandiz ME, Castro-Sanchez AM, Mataran-Penarrocha GA, Guisado-Barrilao R, Garcia-Rios MC, Moreno-Lorenzo C. A randomized controlled trial of a mixed Kinesio taping-compression technique on venous symptoms, pain, peripheral venous flow, clinical severity and overall health status in postmenopausal women with chronic venous insufficiency. Clin Rehabil. 2014 Jan;28(1):69-81. doi: 10.1177/0269215512469120. Epub 2013 Feb 20. PMID 23426563